CLINICAL TRIAL: NCT07160894
Title: Evaluation of Nucleotide-Binding Oligomerization Domain-Containing Protein (NOD) 1 and NOD 2 in Different Periodontal Conditions
Brief Title: Evaluation of Nucleotide-Binding Oligomerization Domain-Containing Protein (NOD) 1 and NOD 2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Melis Yilmaz, Associate Prof Dr, Medipol University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 672
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Periodontal Diseases Inflammation
Keywords: periodontal disease NOD

STUDY DESIGN:
Intervention Model Description: Saliva and serum of periodontitis patients collected for analyzing NOD1, NOD2, IL-10 and IL-6
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator (Active Comparator): Collection of patients' saliva and serum and analysis of sample molecules.
  Interventions: Other: Saliva and Serum sampling
- Experimental (Experimental): ELISA method will be used to evaluate NOD1 and NOD2, IL-10, IL-6 molecules in the saliva and serum samples obtained.
  Interventions: Other: Saliva and Serum sampling

INTERVENTIONS:
Other: Saliva and Serum sampling — Saliva were collected to analyze the selected markers as unstimulated samples during the early hours of the day. The saliva was centrifuged and then transferred into Eppendorf tubes. Venous puncture was performed after saliva collection and 5 mL of blood samples were collected by qualified staff from each participant.Saliva and serum were then stored at -80 °C until analysis.
Other: Saliva and Serum sampling — ELISA method will be used to measure IL-10 and IL-6 values in collected saliva and serum samples. For ELISA analysis, a commercial kit (Sunred Bio, Shanghai, China) pre-coated with human selected antibodies will be used.

SUMMARY:
The host immune response to microorganisms is primarily recognized by pattern recognition receptors (PRRs), including toll-like receptors and nucleotide-binding oligomeric domain (NOD) receptors (NLRs). The aim of this study was to examine the relationship between periodontal disease and NOD in serum and saliva samples.

DETAILED DESCRIPTION:
Healthy participants (n:25), gingivitis (n:25) patients and stage III, grade B periodontitis (n:25) patients enrolled for this study. Clinical periodontal parameters and salivary flow rate were noted. Serum and saliva samples were collected to measure NOD1, NOD2, IL-10 and IL-6 levels.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy

  * clinical diagnosis of periodontal health
  * clinical diagnosis of periodontitis
  * clinical diagnosis of gingivitis

Exclusion Criteria:

* • history of regular use of systemic antibiotics anti-inflammatory, or antioxidant drugs (previous 3 months)

  * nonsurgical periodontal treatment (previous 6 months)
  * surgical periodontal treatment (previous 12 months)
  * presence of<10 teeth
  * current medications affecting gingival health (calcium channel blockers, phenytoin, cyclosporine, and hormone replacement therapy)
  * diabetes
  * diagnosis of rheumatoid arthritis
  * pregnancy
  * lactating
  * smoking
  * excessive alcohol consumption.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-03-12 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Pocket probing depth | 6 months
  Measurement of the depth of a sulcus or periodontal pocket determined by measuring distance from a gingival margin to the base of the sulcus or pocket with a calibrated periodontal probe.
Clinical attachment level | 6 months
  Clinical attachment level (or loss, CAL) is a more accurate indicator of the periodontal support around a tooth than probing depth alone. CAL is measured from a fixed point on the tooth that does not change, the CEJ.
  To calculate CAL, two measurements are needed: distance from the gingival margin to the CEJ and probing depth.
  In recession: probing depth (+) gingival margin to the CEJ (add). In tissue overgrowth: probing depth (-) gingival margin to the CEJ (subtract)
Bleeding on probing | 6 months
  Referring to bleeding that is induced by gentle manipulation of the tissue at the depth of the gingival sulcus, or interface between the gingiva and a tooth.

SECONDARY OUTCOMES:
Saliva and serum samples processing and analyses | 1 month
  Saliva and serum samples obtained for each patient were used for cytokine analysis. Prepared samples were analyzed for NOD1, NOD2, IL-10 and IL-6 using commercial ELISA kits

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, School of Dentistry, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No